CLINICAL TRIAL: NCT02885376
Title: Phase II Study of Dentoxol® Mouthrinse for Oral Mucositis Secondary to Radiation Therapy for Head and Neck Cancer
Brief Title: Study of Dentoxol® Mouthrinse for Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ingalfarma SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ING-001
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Oral Mucositis
Keywords: Mucositis
MeSH Terms: conditions — Stomatitis; Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dentoxol (Experimental): Dentoxol® is a proprietary mouthrinse that has anti-inflammatory, antimicrobial and analgesic effects. Subjects will use Dentoxol® mouthrinse 5 times each day, starting on the first day of radiation therapy and ending on the last day of radiation therapy.
  Interventions: Device: Dentoxol
- Placebo (Placebo Comparator): The placebo rinse will be identical in color, taste and consistency as the Dentoxol rinse and will be packaged in identical bottles with the same labels. Subjects will use placebo mouthrinse 5 times each day, starting on the first day of radiation therapy and ending on the last day of radiation therapy.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Dentoxol — Mouthrinse
  Arms: Dentoxol
Device: Placebo — Mouthrinse
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of Dentoxol® mouthrinse in reducing the severity of oral mucositis secondary to radiation therapy for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Planned to receive radiation therapy for cancer of the oral cavity, oropharynx, nasopharynx, hypopharynx or larynx, with or without concomitant chemotherapy.
* Planned to receive at least 5000cGy radiation therapy to at least 2 of 12 pre-specified areas in the oral cavity

Exclusion Criteria:

* Unable to give written informed consent
* Known allergy/intolerance to any component of the study rinse or placebo
* Planning to use any contraindicated medications during the study period (pain medications are allowed)
* Age below 18 years
* Pregnant or nursing (If the patient is a woman of childbearing potential, a pregnancy test must be performed within fourteen days before enrollment in the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-11; Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Incidence of severe oral mucositis, defined as grade 3 or 4 on the World Health Organization (WHO) scale | First day of radiation therapy through last day of radiation therapy (5-8 weeks)

SECONDARY OUTCOMES:
Duration of and time to onset of severe oral mucositis, defined as grade 3 or 4 on the World Health Organization (WHO) scale. | First day of radiation therapy through last day of radiation therapy (5-8 weeks)
Mouth pain scores, as measured in the Oral Mucositis Daily Questionnaire (OMDQ). | First day of radiation therapy through last day of radiation therapy (5-8 weeks)
Ability to eat, drink, and swallow, as measured in the Oral Mucositis Daily Questionnaire (OMDQ). | First day of radiation therapy through last day of radiation therapy (5-8 weeks)
Weight loss, as measured by the difference between weight on first and last day of radiation therapy. | First day of radiation therapy through last day of radiation therapy (5-8 weeks)
Use of opioid analgesics for oral mucositis pain, as expressed in morphine equivalents. | First day of radiation therapy through last day of radiation therapy (5-8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastián Sole, Principal Investigator — Clinica IRAM
Locations (3):
- Chile (3):
  - Clinica IRAM, Santiago
  - Fundación Arturo López Pérez, Santiago
  - Instituto Nacional del Cáncer, Santiago

IPD SHARING:
Plan to Share IPD: No